CLINICAL TRIAL: NCT05331456
Title: Alveolar Cleft Repair Using Osteoinductive Ceramics in Children With Unilateral Cleft Lip and Palate
Brief Title: Alveolar Cleft Repair Using Osteoinductive Ceramics
Acronym: ACROSTIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Radboud University Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Academisch Ziekenhuis Groningen (Other); Medisch Centrum Leeuwarden (Unknown)
Responsible Party: Principal Investigator, Nard Janssen, N.G. Janssen, Prinicpal Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL75562.041.21
Record Dates: First submitted 2022-04-11; First posted 2022-04-15 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Cleft Palate Children; Cleft Alveolar Ridge; Cleft Lip and Palate
Keywords: cleft palate; cleft lip; alveolar cleft; calcium phosphate ceramics; bone graft
MeSH Terms: conditions — Cleft Lip; Cleft Palate

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alveolar cleft repair using autologous bone from the mandibular symphysis (Other): Control group
  Interventions: Device: Unilateral alveolar cleft repair
- Alveolar cleft repair using a biphasic clacium phosphate putty (Other): Study group
  Interventions: Device: Unilateral alveolar cleft repair

INTERVENTIONS:
Device: Unilateral alveolar cleft repair — Early secondary alveolar cleft repair is performed in children with a unilateral alveolar cleft using eirther autologous bone or a calcium phosphate based putty

SUMMARY:
In this study, patients with unilateral cleft lip and palate are enrolled in a multicenter stepped wedge randomized trial ithat compares alveolar cleft closure using autologous bone harvested form the mandibular symphysis with an osteoinductive biphasic calcium phosphate putty.

DETAILED DESCRIPTION:
Rationale: Patients who undergo alveolar cleft grafting have to deal with postoperative pain and comorbidity due to harvesting of autologous bone.

Objective: To evaluate if using calcium phosphate based scaffolds for alveolar cleft grafting is as effective as the use of an autologous bone graft.

Study design: A 'stepped wedge' randomized controlled trial will be conducted by four centres.

Study population: Children between the ages of 8 to 12 years with a unilateral alveolar cleft.

Intervention: Study group undergoes alveolar cleft grafting with the use of a calcium phosphate based scaffold, the control group undergoes the same procedure, but with the use of an autologous chin bone graft.

Main study parameters/endpoints: Main study outcome is one year postoperative residual bone volume in the reconstructed alveolar cleft. Secondary objectives of importance are postoperative pain and eruption of the tooth adjacent to the cleft through the reconstructed area.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients in the control group will undergo a procedure that is currently seen as the gold standard. Patients in the study group will undergo the exact same risks as the control group, except there is no risk for donor site morbidity and postoperative pain is significantly less. Postoperative clinical and radiological evaluation of both groups is according to current treatment standards.

ELIGIBILITY:
Inclusion Criteria:

* unilateral alveolar cleft, early secondary alveolar cleft closure

Exclusion Criteria:

* cleft lip and palate in a syndromic context

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Bone volume | 1 year postoperatively
  One year postoperative residual bone volume

SECONDARY OUTCOMES:
Postoperative pain | Day 1 to 7 postoperatively
  Postoperative pain on a 1 to 10 scale
Canine eruption | 1 year postoperatively
  Eruption of the canine (or lateral incisor) adjacent to the alevolar cleft

CONTACTS AND LOCATIONS:
Overall Officials: Nard Janssen, MD, DDS, PhD, Principal Investigator — UMC Utrecht
Locations (4):
- Netherlands (4):
  - Amsterdam UMC, Amsterdam
  - UMC Groningen, Groningen
  - Radboud UMC, Nijmegen
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No